CLINICAL TRIAL: NCT04044001
Title: A Prospective Phase Ib/IIa, Active-controlled, Randomized, Open-label Study to Evaluate the Safety, Tolerability, Extended Early Bactericidal Activity and Pharmacokinetics of Multiple Oral Doses of BTZ-043 Tablets in Subjects With Newly Diagnosed, Uncomplicated, Smear-positive, Drug-susceptible Pulmonary Tuberculosis
Brief Title: BTZ-043 - Multiple Ascending Dose (MAD) to Evaluate Safety, Tolerability and Early Bactericidal Activity (EBA)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michael Hoelscher (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Radboud University Medical Center (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Prof. Dr. Michael Hoelscher, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: PanACEA-BTZ-043-02
Record Dates: First submitted 2019-07-29; First posted 2019-08-02 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Tuberculoses; Other Specified Pulmonary Tuberculosis
Keywords: Tuberculosis, Pulmonary; Randomized Controlled Trial (RCT); BTZ-043; Tuberculosis; Antitubercular Agents; Gram-positive Bacterial Infections; Escalating dose; Drug-sensitive TB; Early Bactericidal Activity (EBA); Drug-drug-interaction; Pharmacokinetics (PK); Safety; Tolerability; Bactericidal Activity
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis; Gram-Positive Bacterial Infections | interventions — 2-(2-methyl-1,4-dioxa-8-azaspiro(4.5)dec-8-yl)-8-nitro-6-(trifluoromethyl)-4H-1,3-benzothiazin-4-one; Isoniazid; Rifampin; Pyrazinamide; Ethambutol; dolutegravir

STUDY DESIGN:
Intervention Model Description: Stage 1: We will enrol patients sequentially in up to 8 cohorts of at least 3 patients to receive BTZ-043 in ascending doses. Patients in the first cohort will receive the lowest dose of 250mg of BTZ-043 for 14 days.
  After each patient in a cohort has completed at least 7 days, a dosing recommendation for the next cohort will be made using the continual reassessment method (CRM) algorithm.
  Stage 2: This will be a parallel group comparison of 4 treatment regimens. Patients will be randomized to receive either one of three doses of BTZ-043 within the therapeutic window defined in stage 1, or the control regimen of daily doses of Rifafour e-275®, adapted to body weight, for 14 days in the ratio 3:3:3:2.
Who Masked: Outcomes Assessor
Masking Description: Laboratory staff, analysing and evaluating the sputum and safety blood samples of the participants will be blinded to the treatment cohort/arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Stage 1 - Cohort 1 (BTZ 250) (Experimental): Patients will receive 1 tablet of BTZ-043 orally once daily, containing 250mg BTZ-043 from Day 1 through to Day 14
  Interventions: Drug: BTZ-043
- Stage 1 - Cohort 2 (BTZ 500) (Experimental): Patients will receive 2 tablets of BTZ-043 orally once daily, each containing 250mg BTZ-043 (500 mg in total) from Day 1 through to Day 14
  Interventions: Drug: BTZ-043
- Stage 1 - Cohort 3 (BTZ 750) (Experimental): Patients will receive 3 tablets of BTZ-043 orally once daily, each containing 250mg BTZ-043 (750 mg in total) from Day 1 through to Day 14
  Interventions: Drug: BTZ-043
- Stage 1 - Cohort 4 (BTZ 1000) (Experimental): Patients will receive 4 tablets of BTZ-043 orally once daily, each containing 250mg BTZ-043 (1000 mg in total) from Day 1 through to Day 14
  Interventions: Drug: BTZ-043
- Stage 1 - Cohort 5 (BTZ 1250) (Experimental): Patients will receive 5 tablets of BTZ-043 orally once daily, each containing 250mg BTZ-043 (1250 mg in total) from Day 1 through to Day 14
  Interventions: Drug: BTZ-043
- Stage 1 - Cohort 6 (BTZ 1500) (Experimental): Patients will receive 6 tablets of BTZ-043 orally once daily, each containing 250mg BTZ-043 (1500 mg in total) from Day 1 through to Day 14
  Interventions: Drug: BTZ-043
- Stage 1 - Cohort 7 (BTZ 1750) (Experimental): Patients will receive 7 tablets of BTZ-043 orally once daily, each containing 250mg BTZ-043 (1750 mg in total) from Day 1 through to Day 14
  Interventions: Drug: BTZ-043
- Stage 1 - Cohort 8 (BTZ 2000) (Experimental): Patients will receive 8 tablets of BTZ-043 orally once daily, each containing 250mg BTZ-043 (2000 total) from Day 1 through to Day 14
  Interventions: Drug: BTZ-043
- Stage 2 - Arm 1 (BTZ high) (Experimental): Patients will receive a higher dose of BTZ-043, that has proven to be safe in stage 1 orally once daily from Day 1 through to Day 14. The dose of BTZ-043 will be determined after review of safety data from stage 1.
  Interventions: Drug: BTZ-043; Drug: Probe Drug Cocktail; Drug: Dolutegravir 50mg Tab
- Stage 2 - Arm 2 (BTZ medium) (Experimental): Patients will receive a medium dose of BTZ-043, that has proven to be safe in stage 1 orally once daily from Day 1 through to Day 14. The dose of BTZ-043 will be determined after review of safety data from stage 1.
  Interventions: Drug: BTZ-043; Drug: Probe Drug Cocktail; Drug: Dolutegravir 50mg Tab
- Stage 2 - Arm 3 (BTZ low) (Experimental): Patients will receive a lower dose of BTZ-043, that has proven to be safe in stage 1 orally once daily from Day 1 through to Day 14. The dose of BTZ-043 will be determined after review of safety data from stage 1.
  Interventions: Drug: BTZ-043; Drug: Probe Drug Cocktail; Drug: Dolutegravir 50mg Tab
- Stage 2 - Arm 4 (control) (Active Comparator): Patients will receive a standard dose of Rifafour e-275® orally once daily according to body weight from Day 1 through to Day 14. Each tablet of Rifafour e-275® contains 150mg rifampicin, 75mg isoniazid, 400mg pyrazinamide and 275mg ethambutol.
  The daily doses will be given to fasting patients, in accordance with South African Guidelines for treatment of TB. The total number of tablets will be based on the body weight at screening:
  * participants weighing 38 - 54 kg: 3 tablets
  * participants weighing 55 - 70 kg: 4 tablets
  * participants weighing >70 kg: 5 tablets
  Interventions: Drug: Rifafour e-275®

INTERVENTIONS:
Drug: BTZ-043 — BTZ-043 (250mg per tablet)
  Arms: Stage 1 - Cohort 1 (BTZ 250); Stage 1 - Cohort 2 (BTZ 500); Stage 1 - Cohort 3 (BTZ 750); Stage 1 - Cohort 4 (BTZ 1000); Stage 1 - Cohort 5 (BTZ 1250); Stage 1 - Cohort 6 (BTZ 1500); Stage 1 - Cohort 7 (BTZ 1750); Stage 1 - Cohort 8 (BTZ 2000); Stage 2 - Arm 1 (BTZ high); Stage 2 - Arm 2 (BTZ medium); Stage 2 - Arm 3 (BTZ low)
Drug: Rifafour e-275® — Rifafour e-275® (150mg rifampicin, 75mg isoniazid, 400mg pyrazinamide, 275 mg ethambutol per tablet)
  Other Names: Isoniazid, Rifampicin, Pyrazinamide, Ethambutol (HRZE)
  Arms: Stage 2 - Arm 4 (control)
Drug: Probe Drug Cocktail — A probe drug cocktail will be given to randomly selected patients after inclusion on Day 1 and on Day 14 once orally. The probe drug cocktail consists of
  * Caffeine: 1 tablet à 150mg
  * Tolbutamide: 1/4 tablet à 500mg
  * Dextromethorphan: 10 ml syrup à 15mg/5ml
  * Midazolam:2 ml solution à 5mg/5ml
  * Digoxin: 2 tablets à 0.25mg
  Arms: Stage 2 - Arm 1 (BTZ high); Stage 2 - Arm 2 (BTZ medium); Stage 2 - Arm 3 (BTZ low)
Drug: Dolutegravir 50mg Tab — 1 tablet à 50mg Dolutegravir will be given to randomly selected patients after inclusion on Day 1 and on Day 14 once orally.
  Other Names: Tivicay®
  Arms: Stage 2 - Arm 1 (BTZ high); Stage 2 - Arm 2 (BTZ medium); Stage 2 - Arm 3 (BTZ low)

SUMMARY:
This is a prospective, open label, two-centre, randomized, controlled, two-stage, phase Ib/IIa study to evaluate the safety, tolerability, PK, drug-drug interaction and bactericidal activity of BTZ-043 administered orally once daily over 14 days to participants with newly diagnosed, uncomplicated, smear-positive, drug-susceptible pulmonary tuberculosis.

The primary objective is to assess the safety and tolerability of BTZ-043 given over 14 days by evaluation of adverse events during treatment and follow-up period in patients with newly diagnosed, uncomplicated, smear-positive, drug-susceptible pulmonary tuberculosis.

DETAILED DESCRIPTION:
This is a prospective, open label, two-centre, randomized, controlled, two-stage, phase Ib/IIa study to evaluate the safety, tolerability, PK, drug-drug interaction and bactericidal activity of BTZ-043 administered orally once daily over 14 days to participants with newly diagnosed, uncomplicated, smear-positive, drug-susceptible pulmonary tuberculosis:

Stage 1 is an escalating dose design in up to eight cohorts receiving different doses of BTZ-043 to define a safe dose corridor for BTZ-043. The focus of this stage is on adverse events, PK and a food-effect PK-evaluation .

Stage 2 is a parallel group comparison of 4 arms receiving different treatment regimens: three arms to receive BTZ-043 in different doses within the safe corridor defined in stage 1, compared to one arm receiving Rifampicin, Isoniazid, Pyrazinamide, and Ethambutol as a control. This stage is focusing on adverse effects, early bactericidal activity (EBA), PK and an evaluation of PK drug-drug interaction potential.

A total of up to 77 male and female patients, aged ≥ 18 - 64 years, with newly diagnosed, smear positive, drug sensitive pulmonary tuberculosis will be enrolled.

Allocation of patients will be carried out in two stages:

Stage 1: for each cohort 3 patients will be enrolled, treated and followed-up accordingly, starting with cohort 1. In a Trial Steering Committee (TSC) meeting, decision will be made on the dose in the next cohort.

Dose escalation steps to be followed, if no safety concerns arise:

* Cohort 1: patients to receive 250 mg BTZ-043
* Cohort 2: patients to receive 500 mg BTZ-043
* Cohort 3: patients to receive 750 mg BTZ-043
* Cohort 4: patients to receive 1000 mg BTZ-043
* Cohort 5: patients to receive 1250 mg BTZ-043
* Cohort 6: patients to receive 1500 mg BTZ-043
* Cohort 7: patients to receive 1750 mg BTZ-043
* Cohort 8: patients to receive 2000 mg BTZ-043

Patients receiving the investigational drug in cohorts 1 - 8 will take BTZ-043 in fasting state for 13 days and after a pre-defined high-fat, high-caloric meal on day 14.

After all patients of a current cohort have completed at least 7 days of dosing, the TSC, composed of the national principal investigator (PI), the trial statistician, the sponsor representative and two independent scientists, will review safety data, including clinical, lab and electrocardiography (ECG) data, to assess whether dose limiting toxicity of BTZ-043, as defined below, has been observed in any participant. Depending on the outcome, the TSC will then decide on dose escalation, or on enrolling more participants to the same or a lower dose in the following cohort, according to dose escalation and stopping rules.

After the end of stage 1, the TSC will decide which of the BTZ-043 doses, which are deemed to not exceed the acceptable toxicity level, are to be moved to stage 2.

Stage 2: after the highest possible dose of the investigational drug, that has proven to be safe within the 1st stage, is identified, all remaining patients will be recruited and randomised to receive one of three different doses of BTZ-043 or to control treatment with Rifafour e-275® at a ratio of 3:3:3:2 favouring the experimental treatment.

Stage 2 is focusing on adverse effects, early bactericidal activity (EBA), PK and an evaluation of PK drug-drug interaction potential.

Allocation of patients:

* Arm 1: patients to receive BTZ-043 in a higher dose
* Arm 2: patients to receive BTZ-043 in a medium dose
* Arm 3: patients to receive BTZ-043 in a lower dose
* Control Arm 4: patients to receive Rifafour e-275® as control treatment

Participants will take in BTZ-043 in either fasted or fed state, depending on which state has shown to lead to higher exposure during the 1st stage.

Additional measurements in the 2nd stage in BTZ-arms 1 to 3 only:

• Drug-drug interactions will be investigated: patients, who have been randomized to BTZ-043 arms, will additionally be randomized to receive either a probe drug cocktail, with drugs specifically metabolized by certain enzymes, or dolutegravir at a ratio of 2:1. Probe drugs or Dolutegravir (DTG) will be given pre-BTZ on day 0 and on day 14.

After the course of study drugs is completed (on day 14), all patients (in stage 1 and stage 2) will be referred to a government clinic to complete their course of tuberculosis (TB) according to national standards for a total of 6 months of first-line therapy.

ELIGIBILITY:
General inclusion criteria:

1. Provide written, informed consent prior to all trial-related procedures including HIV testing.
2. Understand and willing to comply with the study procedures.
3. Male or female adults, aged 18 up to and including 64 years.
4. Body weight ≥ 40 kg.
5. Participants are either unable to conceive/father children AND/OR they will be using two effective methods of contraception, including methods used by the patient's sexual partner(s). At least one to be a barrier method.

   Disease-specific inclusion criteria:
6. Newly diagnosed, previously untreated, drug-susceptible pulmonary TB
7. Chest X-ray which is consistent with TB
8. Ability to produce an adequate volume of sputum (at least 10ml estimated overnight production)
9. ≥ 1 sputum sample from concentrated sputum positive for acid-fast bacilli on microscopy (at least 1+ on the International Union Against Tuberculosis and Lung Disease/World Health Organization (IUATLD/WHO) scale) from either a spot sputum or overnight sputum sample.

General exclusion criteria:

1. Poor general condition, where delay in treatment cannot be tolerated or death within three months is likely, as assessed by the investigator.
2. The patient is pregnant or breast-feeding.

   Disease-specific exclusion criteria:
3. The patient is infected with HIV.
4. The patient has a known intolerance to any of the study drugs or concomitant disorders or conditions for which study drugs or standard TB treatment are contraindicated.
5. Treatment with any other investigational drug within 1 month prior to enrolment or enrolment into other clinical (intervention) trials during participation.
6. The patient has a history of or current evidence of clinically relevant cardiovascular metabolic, gastrointestinal, neurological, psychiatric or endocrine diseases, malignancy or any other condition, that will influence treatment response, study adherence or survival in the judgement of the investigator, especially:

   1. Clinically significant evidence of severe TB (e.g. miliary TB, TB meningitis, excluding limited lymph node involvement)
   2. Serious lung conditions other than TB or significant respiratory impairment in the discretion of the investigator
   3. Neuropathy, epilepsy or significant psychiatric disorder
   4. Any diabetes mellitus
   5. Cardiovascular disease, such as myocardial infarction, heart failure, coronary heart disease, arrhythmia, tachyarrhythmia, or pulmonary hypertension
   6. Current or history of hypertension (systolic blood pressure >135 mmHg and/or diastolic blood pressure of >85 mmHg) AND/OR ever received antihypertensive treatment)
   7. Long QT syndrome or family history of long QT syndrome or sudden death of unknown or cardiac-related cause
   8. Alcohol or other drug abuse, that is sufficient to significantly compromise the safety or cooperation of the patient, includes substances prohibited by the protocol, or has led to significant organ damage, at the discretion of the investigator

   Laboratory exclusion criteria at screening:
7. Serum amino aspartate transferase (AST) and/or alanine aminotransferase (ALT) activity >2x the upper limit of normal (ULN)
8. serum alkaline phosphatase (ALP) or y-glutamyl transferase (GGT) > 2x the ULN
9. serum total bilirubin level >1.5 times the ULN
10. estimated creatinine clearance (eCrCl) using the Cockcroft and Gault formula level lower than 60 mls/min
11. haemoglobin level <8.0 g/dL
12. platelet count <100,000/mm3
13. serum potassium below the lower level of normal (LLN) for the laboratory

    ECG-specific exclusion criteria:
14. corrected QT interval (QTc)F of > 450 milliseconds (ms)
15. Atrioventricular (AV) block with PR interval > 200 ms
16. QRS complex > 120 ms
17. any other changes in the ECG that are clinically relevant as per discretion of the investigator

    Restricted medication:
18. Treatment with drugs active against Mycobacterium Tuberculosis (MTB) within the last 3 months prior to screening
19. Requires medication as included in the following drug classes within 2 weeks prior to the first dose of study treatment:

    * medication that prolongs the QTc interval
    * Cytochrome P450 (CYP450) inhibitors or inducers, including grapefruit containing foods / beverages and St. John's Wort
    * Antacids or antipeptic drugs (antacids, H2 blockers, proton pump inhibitors)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of BTZ-043 | Day 1 to Day 22
  Safety and tolerability of BTZ-043 will be assessed by evaluation of Adverse Events (AEs) during treatment- and follow-up phase

SECONDARY OUTCOMES:
Bactericidal Activity Endpoint - MGIT | Day -1 to Day 14
  • changes in time to detection in the Mycobacteria Growth Indicator Tube (MGIT™) liquid media culture system from baseline
Bactericidal Activity Endpoint - CFU | Day -1 to Day 14
  • changes in solid media colony forming units (CFU) from baseline
Bactericidal Activity Endpoint - LAM | Day -1 to Day 14
  • changes in sputum lipoarabinomannan (LAM) concentration from baseline
Bactericidal Activity Endpoint - MBLA | Day -1 to Day 14
  • changes in sputum molecular bacterial load assay (MBLA) from baseline
Pharmacokinetic Endpoint - BTZ-043 - AUC | Day 1, 12 and 14
  The PK of BTZ-043 and its two major metabolites BTZ-045S and M2 after a single dose and at steady state will be evaluated by measuring the area under the plasma concentration curve (AUC)
Pharmacokinetic Endpoint - BTZ-043 - Cmax | Day 1, 12 and 14
  The PK of BTZ-043 and its two major metabolites BTZ-045S and M2 after a single dose and at steady state will be evaluated by measuring the observed maximum concentration (Cmax)
Pharmacokinetic Endpoint - BTZ-043 - Tmax | Day 1, 12 and 14
  The PK of BTZ-043 and its two major metabolites BTZ-045S and M2 after a single dose and at steady state will be evaluated by measuring the time to reach Cmax (Tmax)
Pharmacokinetic Endpoint - BTZ-043 - Cmin | Day 1, 12 and 14
  The PK of BTZ-043 and its two major metabolites BTZ-045S and M2 after a single dose and at steady state will be evaluated by measuring the minimum observed plasma concentration 24 hours following the last dose (Cmin)
Pharmacokinetic Endpoint - BTZ-043 - Cl | Day 1, 12 and 14
  The PK of BTZ-043 and its two major metabolites BTZ-045S and M2 after a single dose and at steady state will be evaluated by measuring the Clearance (Cl)
Pharmacokinetic Endpoint - BTZ-043 - Vd | Day 1, 12 and 14
  The PK of BTZ-043 and its two major metabolites BTZ-045S and M2 after a single dose and at steady state will be evaluated by measuring the Volume of distribution (Vd)
Pharmacokinetic Endpoint - BTZ-043 - T1/2 | Day 1, 12 and 14
  The PK of BTZ-043 and its two major metabolites BTZ-045S and M2 after a single dose and at steady state will be evaluated by measuring the Elimination half-life (T1/2)
Pharmacokinetic Endpoint - BTZ-043 - pharmacodynamics (PD) | Day 1, 12 and 14
  The PK of BTZ-043 and its two major metabolites BTZ-045S and M2 after a single dose and at steady state will be evaluated by measuring the Relation of efficacy measurements to pharmacokinetic indices of BTZ-043 and its metabolites (AUC, Cmax)
Pharmacokinetic Endpoint - Population PK AUC | Day 1, 12 and 14
  A population PK-analysis of BTZ-043 and its two major metabolites will be carried out by measuring the AUC and describing PK differences of BTZ-043 and its main metabolites between subjects to quantify inter-individual variability, suitable for evaluation of alternative dosing regimens
Pharmacokinetic Endpoint - Population PK Cmax | Day 1, 12 and 14
  A population PK-analysis of BTZ-043 and its two major metabolites will be carried out by measuring the Cmax and describing PK differences of BTZ-043 and its main metabolites between subjects to quantify inter-individual variability, suitable for evaluation of alternative dosing regimens
Pharmacokinetic Endpoint - Food Effect PK AUC | Day 14
  The effect of food on the exposure of the BTZ-043 and its two major metabolites will be determined by measuring the AUC of BTZ-043 and its main metabolites and by evaluating the change after a high fat high calorie meal in comparison to the AUC under fasting conditions during the 1st stage.
Pharmacokinetic Endpoint - Food Effect PK Cmax | Day 14
  The effect of food on the exposure of the BTZ-043 and its two major metabolites will be determined by measuring the Cmax of BTZ-043 and its main metabolites and by evaluating the change after a high fat high calorie meal in comparison to the Cmax under fasting conditions during the 1st stage.
Pharmacokinetic Endpoint - Probe Drugs PK AUC | Day 0 and 14
  The effect on BTZ-043 at steady state on hepatic enzyme and P-glycoprotein activity (induction vs. inhibition) will be evaluated by measuring changes in AUC of the probe drugs administered on day 0, and day 14 during the 2nd stage.
Pharmacokinetic Endpoint - Probe Drugs PK Cmax | Day 0 and 14
  The effect on BTZ-043 at steady state on hepatic enzyme and P-glycoprotein activity (induction vs. inhibition) will be evaluated by measuring changes in Cmax of the probe drugs administered on day 0, and day 14 during the 2nd stage.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoelscher, Prof, Study Director — University Hospital, LMU Munich, Division of Infectious Diseases and Tropical Medicine; Andreas Diacon, Prof, Principal Investigator — TASK Applied Science Clinical Research Centre
Locations (2):
- South Africa (2):
  - TASK Applied Sciences Clinical Research Centre, Cape Town
  - University of Cape Town Lung Institute (UCTLI), Cape Town

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heinrich N, de Jager V, Dreisbach J, Gross-Demel P, Schultz S, Gerbach S, Kloss F, Dawson R, Narunsky K, Matt L, Wildner L, McHugh TD, Fuhr U, Aldana BH, Mouhdad C, Brake LT, Boeree MJ, Aarnoutse RE, Svensson EM, Gong X, P J Phillips P, Diacon AH, Hoelscher M; PanACEA-TB consortium. Safety, bactericidal activity, and pharmacokinetics of the antituberculosis drug candidate BTZ-043 in South Africa (PanACEA-BTZ-043-02): an open-label, dose-expansion, randomised, controlled, phase 1b/2a trial. Lancet Microbe. 2025 Feb;6(2):100952. doi: 10.1016/j.lanmic.2024.07.015. Epub 2025 Jan 7. PMID 39793592